CLINICAL TRIAL: NCT06338761
Title: Prognostic Impact of Switching to E-Cigarette Use in Smokers With Coronary Artery Disease Following Percutaneous Coronary Intervention: A Nationwide Cohort Study
Brief Title: Switching to E-cigarette After PCI
Acronym: E-cig-PCI
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ki Hong Choi, Professor, Samsung Medical Center
Other Study IDs: E-cigarette PCI
Record Dates: First submitted 2024-03-24; First posted 2024-04-01 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous coronary intervention; E-cigarette; Smoking
MeSH Terms: conditions — Coronary Artery Disease; Vaping; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Continued combustible cigarette use: continued combustible cigarettes users after PCI
- Switching to E-cigarette: switching to E-cigarette users after PCI
  Interventions: Behavioral: Switching to E-cigarette
- Quitter: quitters after PCI
  Interventions: Behavioral: Smoking cessation

INTERVENTIONS:
Behavioral: Smoking cessation — Stop smoking
  Groups: Quitter
Behavioral: Switching to E-cigarette — Switching to E-cigarette
  Groups: Switching to E-cigarette

SUMMARY:
Despite the increasing popularity of electronic cigarettes (E-cigarettes), the prognostic impact of switching to E-cigarettes in smokers with coronary artery disease (CAD) who underwent percutaneous coronary intervention (PCI) remains uncertain.

DETAILED DESCRIPTION:
Recently, several studies have reported that, although lower than combustible cigarette users, E-cigarette users had a significantly higher risk of future myocardial infarction (MI) or cardiovascular disease compared with non-smokers or quitters. However, because all previous studies has focused on the general healthy population, these results cannot be extrapolated for patients who already proven atherosclerotic cardiovascular disease (ASCVD), such as undergoing percutaneous coronary intervention (PCI) for coronary artery disease (CAD). Although Busch et al. previously reported that a significant minority of patients are using E-cigarettes post-acute coronary syndrome smokers, a paucity of data exists regarding the impact of such transitions on clinical outcomes in current smoker patients with CAD who have undergone PCI. In light of these considerations, the current study sought to address this gap in knowledge by evaluating the prognostic implications of smoking habit changes, including E-cigarette use, among CAD patients with current smoking status following PCI.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent health screening 3 years before and after the PCI

Exclusion Criteria:

* history of cancer
* history of ischemic stroke
* died within the first 3 months of follow-up from the index date
* Newly developed acute MI or received additional PCI or CABG from the index PCI date to the study index date

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with coronary artery disease who underwent health screening 3 years before and after the PCI
Sampling Method: Non-Probability Sample
Enrollment: 17973 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
MACE | 5 years after PCI
  Major adverse cardiac event

SECONDARY OUTCOMES:
Cardiovascular death | 5 years after PCI
  death from cardiovascular cause
All-cause death | 5 years after PCI
  death from any cause
Spontaneous myocardial infarction | 5 years after PCI
  MI with hospitalization
Repeat revascularization | 5 years after PCI
  additional PCI or CABG

CONTACTS AND LOCATIONS:
Overall Officials: Ki Hong Choi, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kang D, Choi KH, Kim H, Park H, Heo J, Park TK, Lee JM, Cho J, Yang JH, Hahn JY, Choi SH, Gwon HC, Song YB. Prognosis after switching to electronic cigarettes following percutaneous coronary intervention: a Korean nationwide study. Eur Heart J. 2025 Jan 3;46(1):84-95. doi: 10.1093/eurheartj/ehae705. PMID 39429032